CLINICAL TRIAL: NCT03510351
Title: Clinical Outcomes With Ceftolozane-tazobactam in Patients With Multi Drug Resistant (MDR) Pseudomonas Aeruginosa Infections
Brief Title: Clinical Outcomes With Ceftolozane-tazobactam for MDR Pseudomonas Infections
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Temple University (Other)
Responsible Party: Sponsor
Other Study IDs: Gallagher
Record Dates: First submitted 2017-11-27; First posted 2018-04-27 (Actual); Last update posted 2018-04-27 (Actual); Status verified 2018-04

CONDITIONS: Pseudomonas Infections; Pseudomonas Aeruginosa
MeSH Terms: conditions — Pseudomonas Infections | interventions — ceftolozane, tazobactam drug combination

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Treated subjects: All patients with Pseudomonas infections treated with ceftolozane-taezobactam who meet the inclusion criteria
  Interventions: Drug: Ceftolozane-Tazobactam

INTERVENTIONS:
Drug: Ceftolozane-Tazobactam — Subjects treated with ceftolozane-tazobactam for Pseudomonas infections

SUMMARY:
This study will describe clinical outcomes in patients who received ceftolozane-tazobactam for a Pseudomonas aeruginosa infection. Primary outcomes include 30-day and in-hospital mortality.

DETAILED DESCRIPTION:
Very little data is available to evaluate the use of ceftolozane-tazobactam in MDR Pseudomonas aeruginosa infections. Additionally, there is currently no standard recommendation for the treatment of MDR Pseudomonas aeruginosa infections, and multiple agents are often used in combination which increases the probability of adverse effects in addition to leading to possibly more resistance and higher costs of care. This is particularly relevant since the primary alternative drugs for MDR Pseusomonas aeruginosa infections are aminoglycosides and polymyxins, two categories of agents with significant adverse effects and suboptimal pharmacokinetics that limit efficacy.

This is a multicenter study designed to collect retrospective data on clinical outcomes of patients treated with ceftolozane-tazobactam in the hospital. The primary outcomes include 30-day and in-hospital mortality. Microbiological and clinical cure will be assessed as secondary outcomes. Microbiological outcomes will be defined as: cure- a repeat culture was negative; failure- repeat cultures were not negative or the patient died before repeat cultures could be obtained; presumed cure- repeat cultures were not taken but clinical cure occurred. Clinical outcomes will be defined as: clinical success- signs and symptoms o the index infection resolved at the end of therapy; clinical failure- signed and symptoms remained at the end of therapy or the patient died; indeterminate- it was not possible to determine the clinical outcome at the end of therapy.

Patient information will be collected from Temple University Hospital as well as 20 other hospital sites. The source population will be all adult patients who received ceftolozane-tazobactam for greater than 24 hours in each of the hospital sites between December 19, 2014 and December 31, 2016. Participating hospital sites will review clinical charts to identify and enroll a target of 5-15 subjects per site. We have a targeted enrollment of 200 subjects. All involved parties will use the Research Electronic Data Capture (RedCap) database based at Temple University for data collection and storage.

We will be utilizing existing electronic data and will have no direct contact with or recruit research subjects. Because this is a study with retrospective data collection, enrolled patients will have received treatment as determined by the treating physicians in accordance with standard of care. To limit bias in the selection of subjects, investigators will be asked to identify and consecutively enroll all eligible patients treated with ceftolozane-tazobactam within the study period.

ELIGIBILITY:
Inclusion Criteria:

* Greater than 18 years old
* Cultures positive Pseudomonas aeruginosa from any source
* Received ceftolozane-tazobactam for at least 24 hrs

Exclusion Criteria:

* Protected populations
* Prisoners, pregnant women, children

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who had Pseudomonas aeruginosa infection and received ceftolozane-tazobactam for at least 24 hrs for treatment.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2019-02-28 (Estimated); Study Completion 2019-02-28 (Estimated)

PRIMARY OUTCOMES:
Mortality | 30 days
  30-day mortality

SECONDARY OUTCOMES:
Microbiological cure | Up to 12 weeks
  Negative repeated bacterial cultures collected from site of infection

CONTACTS AND LOCATIONS:
Overall Officials: Peter Doukas, Ph.D, Study Chair — Temple University - School of Pharmacy
Locations (1):
- Temple University, School of Pharmacy, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No